CLINICAL TRIAL: NCT02687594
Title: Non-interventional Study to Investigate the Short and Long Term Real-life Safety, Effectiveness, and Adherence of Velphoro® in Patients With Hyperphosphataemia Undergoing Haemodialysis or Peritoneal Dialysis
Brief Title: Non-interventional Study to Investigate the Short and Long Term Real-life Safety, Effectiveness, and Adherence of Velphoro® in Patients With Hyperphosphataemia Undergoing Haemodialysis (HD) or Peritoneal Dialysis (PD)
Acronym: VERIFIE
Status: Completed | Type: Observational
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: VFMCRP-MEAF-PA21-01-EU
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — sucroferric oxyhydroxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- single group: sucroferric oxyhydroxide
  Interventions: Drug: sucroferric oxyhydroxide

INTERVENTIONS:
Drug: sucroferric oxyhydroxide — The non-interventional design allows the observation of patients in a broad range of settings reflecting routine clinical practice. All decisions on therapeutic or diagnostic procedures, treatments, management of the disease, or resource utilisation will be at the full discretion of the treating physician without interference by a sponsor or study protocol. All treatment decisions will follow the real-life treatment behaviour.
  Other Names: PA21 (Velphoro)

SUMMARY:
An oral highly potent P binder Velphoro is a mixture of polynuclear iron(III) oxyhydroxide, sucrose, and starches. It was well tolerated in the clinical development program. The approved indication in the European Union (EU) is to control serums phosphorus (sP) levels in adult CKD (Chronic kidney disease) patients on HD (Haemodialysis) or PD (Peritoneal dialysis).

It is of major interest to observe the drug in daily use outside of controlled trial settings. The Marketing Authorisation Holder wishes to obtain further systematic data within a non-interventional study to investigate short and long-term safety.

Effectiveness and Treatment adherence during real-life use will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Signed informed consent
* Indication for Velphoro treatment in accordance with the SmPC
* Prevalent dialysis patients with a dialysis vintage of at least 6 months (HD or PD)
* Treatment-naïve or pre-treated with anti-hyperphosphataemic therapy

Exclusion Criteria:

* Prior participation in this NIS (Non-Interventional Study)
* Parallel participation in an interventional study
* Enrolment in a prior clinical trial with Velphoro

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients with a diagnosis of hyperphosphataemia who are due to be treated with Velphoro according to the product's Summary of Product Characteristics (SmPC) are eligible for this non-interventional study.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-04-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Drug Reactions (ADRs) | through study completion, up to 42 months
Proportion of Adverse Drug Reactions (ADRs) | through study completion, up to 42 months

SECONDARY OUTCOMES:
Patient Reported Outcome questionnaire - Adherence to Velphoro based on the standard Morisky questionnaire | through study completion, up to 42 months
  Patient reported outcomes will be evaluated by descriptive statistics
Patient Reported Outcome questionnaire - Perceived Pill based on the ACTG questionnaire | through study completion, up to 42 months
  Patient reported outcomes will be evaluated by descriptive statistics
Patient Reported Outcome questionnaire - Treatment satisfaction based on the 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) | through study completion, up to 42 months
  Patient reported outcomes will be evaluated by descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Walpen, Dr., Study Chair — Vifor Fresenius Medical Care Renal Pharma
Locations (7):
- Centre Hospitalier LYON-SUD, Pierre-Bénite, France
- Klinikum Coburg, Coburg, Germany
- General Hospital of Athens Laiko, Athens, Greece
- Ospedale Maggiore Policlinico, Milan, Italy
- VU University Medical Center, Amsterdam, Netherlands
- Hospital Universitario Marqués de Valdecilla, Santander, Spain
- Salford Royal Hospitals NHS Trust, Manchester, United Kingdom